CLINICAL TRIAL: NCT02672007
Title: Methods for the Measurement of Respiratory Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Niels Egholm Pedersen, MD, PhD student, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: CAMES-16-001
Record Dates: First submitted 2016-01-11; First posted 2016-02-03 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Rate Measurement Methods.
Keywords: Respiratory rate measurement methods.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Included patients (Other): All included patients will have respiratory rates measured by a research assistant using a criterion standard approach, by the SensiumVitals device and by the ward staff.
  Interventions: Device: SensiumVitals

INTERVENTIONS:
Device: SensiumVitals — The patients will have their respiratory rates, heart rates and temperature (axilla) measured continuously by the SensiumVitals patch.

SUMMARY:
This study aims to investigate these research questions:

1. Is there a difference in the results obtained, when respiratory rate is measured automatically by an electronic device (SensiumVitals® system, Sensium Healthcare) compared with a research assistant using a criterion standard approach?
2. Is there a difference in the results obtained, when respiratory rate is measured automatically by an electronic device (SensiumVitals® system, Sensium Healthcare) compared with hospital staff's current clinical practice?

DETAILED DESCRIPTION:
Respiratory rate is among the first vital signs to change when a deterioration in patient conditions occurs, and that it is highly useful in identifying high-risk patients, patients in pain, risk of death in patients treated for myocardial infarctions and medical patients at risk of cardiac arrest.

Respiratory rate is one of the seven physiological parameters included in the Early Warning Score (EWS), an aggregated track- and trigger-system for risk-stratification of patients in hospital wards at risk of imminent clinical deterioration. EWS includes an escalation protocol, defining when it is necessary for the ward staff to call for assistance and when vital parameters should be measured again.

Manual measurement of respiratory rates is the standard in hospital wards in the Capital Region of Denmark. During the measurement of respiratory rate, patients ideally have to lie still and refrain from talking. This poses a difficulty in daily, clinical practice. Several studies in hospital wards both using and not using an EWS-system report that respiratory rate is often omitted when vital signs are measured.

Even if the respiratory rate is measured regularly, poor inter-observer agreement and reproducibility of measured respiratory rates have been found. Respiratory rates recorded by nurses have been reported to be generally higher than those measured by observers using a standardised approach.

The EWS currently in use is validated using measurements obtained by normal nursing practise. If there is an element of human influence on the measurement of respiratory rate, automation could affect the prognostic properties of EWS in an unpredictable way, even if the automatically measured respiratory rates more reliably reflect the patients' physiology than current clinical practise.

If a systematic difference between the recordings by staff and the electronic devices currently on the market exists, this could have an implication on the EWS scores and subsequently, escalation protocols for patients with elevated EWS could be affected. If this is the case, EWS might even have to be re-validated using machine-measured respiratory rates.

Thus, even as there could be a number of advantages of automating the measurements of respiratory rates in hospital wards, due considerations are required before ward staff's manual measurement of respiratory rate can be replaced by measurements obtained from electronic devices. The purpose of this study is to evaluate if there is a systematic difference in the respiratory rate measurements performed by an electronic device (SensiumVitals® system, Sensium Healthcare) compared with the measurements performed by a research assistant using a criterion standard approach and the ward staff's usual measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Able and willing to give informed consent to participation in the study and necessary data collection.
* Admitted to the general medical short-time ward and planned stay there at the time of inclusion greater than two hours.

Exclusion Criteria:

* Wounds, burns or other conditions that prevent proper attachment of the measurement device, or where wearing the device might cause or increase discomfort from wearing the device.
* Allergies to medical graded tape or ECG electrodes.
* Patients with cardiac pacemaker or implanted defibrillator.
* Any condition or situation preventing proper information, consent and enrolment.
* Respiratory rate measurements by another device using impedance pneumography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Difference in respiratory rate recorded by the research assistant using a criterion standard approach and the SensiumVitals device | 24 Hours
  After enrolment at the general, medical short-time ward a research assistant will measure the patient's respiratory rate using a criterion standard approach. The time of this measurement will be registered, and the corresponding measurement made by the SensiumVitals device will be extracted and used for the comparison. Reported with Bland-Altman plots.

SECONDARY OUTCOMES:
Difference in respiratory rate recorded by the ward staff using standard clinical practice and the SensiumVitals device | 24 Hours
  The ward staff's first measurement of respiratory rate after the patient is enrolled in the study at the general, medical short-time ward as registered in the electronic patient journal. The time of this measurement will be registered, and the corresponding measurement made by the SensiumVitals device will be extracted and used for the comparison. Reported with Bland-Altman plots.

OTHER OUTCOMES:
Early Warning Score recorded by the research assistant | 24 Hours
  Early Warning Score (point score) will be recorded using standard practice by the research assistant. Parameters included in the Early Warning Score: Peripheal arterial oxygen satuation (%), pulse (beats per minute), use of supplementary oxygen (liters per minute), systolic and diastolic blood pressure (mmHg), level of consciousness (AVPU-scale), temperature (degrees celcius) and pulse regularity (yes/no).
Early Warning Score recorded by the ward staff | 24 Hours
  Early Warning Score (point score) recorded using standard practice by the ward staff. Early Warning Score consists of: Peripheal arterial oxygen satuation (%), pulse (beats per minute), use of supplementary oxygen (liters per minute), systolic and diastolic blood pressure (mmHg), level of consciousness (AVPU-scale) and temperature (degrees celcius).

CONTACTS AND LOCATIONS:
Overall Officials: Niels E Pedersen, MD, Principal Investigator — Copenhagen Academy for Medical Education and Simulation, Herlev Hospital, Center for HR, Capital Region of Denmark
Locations (1):
- Copenhagen Academy for Medical Education and Simulation and Medical-Short Time Ward, Herlev Hospital, Herlev, Herlev, Denmark